CLINICAL TRIAL: NCT03120910
Title: Validation of PVI as a Parameter to Predict Fluid Responsiveness
Brief Title: Pleth Variability Index (PVI) to Predict Fluid Responsiveness
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FLEM0005; NCT03075150 (obsolete NCT alias)
Record Dates: First submitted 2017-04-14; First posted 2017-04-19 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Test Subjects (Experimental): All subjects are enrolled into this arm and will receive an investigational pulse CO-Oximeter sensor, including nasal sensors, with the same or similar technology and materials as the Masimo FDA cleared devices and sensors.
  Interventions: Device: Pulse CO-Oximeter Sensor

INTERVENTIONS:
Device: Pulse CO-Oximeter Sensor — Investigational Pulse Oximeter Sensor will measure hemoglobin (SpHb), pulse rate (PR), perfusion index (PI), pleth variability index (PVI), oxygen reserve index (ORI), etc.

SUMMARY:
Interventional data collection study to evaluate the ability of pleth variability index (PVI) to predict fluid responsiveness in comparison with other dynamic parameters including pulse pressure variation (PPV) and stroke volume variation (SVV).

DETAILED DESCRIPTION:
No subjects were enrolled into the validation portion of this study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Scheduled for elective surgery requiring general anesthesia and mechanical ventilation
* Arterial line and Swan-Ganz catheter placement indicated as part of the scheduled surgical procedure

Exclusion Criteria:

* Patients with surgeries at or around site of sensor placement or skin abnormalities affecting the sensor placement area such as psoriasis, eczema, angioma, scar tissue, burn, fungal infection, substantial skin breakdown, nail polish, or acrylic nails that would prevent monitoring of pulse-oximeter physiological parameters during the study
* Patients with cardiac arrhythmias
* Patients with intracardiac shunts

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2018-02-09 (Actual); Study Completion 2018-02-09 (Actual)

PRIMARY OUTCOMES:
Clinical utility of PVI | 1-5 hours
  Correlation between PVI and SVV to assess PVI as a predictor for fluid responsiveness.

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No